CLINICAL TRIAL: NCT07293624
Title: Effects of the Dietary Inflammatory Index on Systemic Inflammation Markers and Gastrointestinal Symptoms in Individuals With Bariatric Surgery
Status: Enrolling by invitation | Type: Observational
Sponsor: Istanbul Bilgi University (Other)
Responsible Party: Principal Investigator, Hande Seven Avuk, Assistant Professor, Head of Nutrition and Dietetic Department, Istanbul Bilgi University
Other Study IDs: BARINFLAMMATION
Record Dates: First submitted 2025-12-07; First posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Bariatric Surgery; Bariatric Sleeve Gastrectomy; Inflamation; Systemic Inflammation; Dietary Inflammatory Index (DII); Systemic Inflammation Markers
Keywords: sleeve gastrectomy; diatary inflammation; bariatric surgery; systemic inflammation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Observational Intervention — This is cross sectional observational study.
Other: Observetional — This is cross-sectional study. Questionnaire, Dietary Inflammatory Index (DII), systemic inflammatory markers, and gastrointestinal symptoms will be investigated.

SUMMARY:
The goal of this observational cross-sectional study is to evaluate the relationships between the Dietary Inflammatory Index (DII), systemic inflammatory markers, and gastrointestinal symptoms in adults aged 18-65 who have undergone bariatric surgery.

The main questions it aims to answer are:

Does the inflammatory potential of the diet affect systemic inflammation levels (such as SII, CRP, and WBC) in the post-operative period?

Is there an association between the DII score and gastrointestinal symptoms (e.g., bloating, gas, abdominal pain)?

Participants who are at least three months post-bariatric surgery will provide dietary intake data to calculate DII scores, undergo blood tests to measure inflammatory markers, and complete assessments regarding their gastrointestinal symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Adult individuals between the ages of 18 and 65,
* Having undergone bariatric surgery at least 3 months prior,
* Individuals who agreed to participate voluntarily in the study and signed the informed consent form,
* Having the cognitive ability/literacy to completely complete the food consumption record and questionnaire forms,
* Individuals with no health conditions that would prevent blood tests,
* Individuals who were regularly followed up after surgery and had no postoperative complications.

Exclusion Criteria:

* Individuals diagnosed with gastrointestinal diseases such as inflammatory bowel disease, celiac disease, or short bowel syndrome before or after bariatric surgery,
* Those with a history of diseases that could affect systemic inflammation, such as autoimmune disease, active infection, or cancer,
* Individuals regularly taking medications that could affect inflammation levels, such as corticosteroids, immunosuppressants, or anti-inflammatory drugs,
* Individuals actively or recently using probiotic supplements,
* Pregnant or breastfeeding women,
* Those with a history of chronic alcohol use or substance abuse,
* Individuals who experienced serious postoperative complications after surgery (e.g., anastomotic leak, serious infection, or conditions requiring reoperation),
* Individuals with cognitive or communication disabilities that prevented them from providing the necessary information and data to the study or who were lost to follow-up,
* Individuals with chronic organ failure,
* Individuals with a psychiatric diagnosis,
* Individuals who did not consent to their data being used for scientific purposes.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Aktif International Uskudar Hospital, Istanbul, Türkiye.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Biochemical Measurements - Fasting blood glucose | at the beginning the study 1 times
  Fasting blood sugar (mg/dL) will be analyzed in the hospital biochemistry laboratory using routine methods from blood samples taken by a nurse at the beginning of the study.
Biochemical Measurement - Lipid Profile | at the beginning the study 1 times
  Participants' biochemical tests (total cholesterol, HDL cholesterol, LDL cholesterol, triglyceride, (mg/dL) will be analyzed in the hospital biochemistry laboratory using routine methods at the beginning of the study from blood samples taken by a nurse after at least 12 hours of fasting and without consuming alcohol for 24 hours before.
Biochemical Measurements - Liver Enzymes | at the beginning the study 1 times
  Participants' liver enzymes tests (ALT, AST, and ALP) (IU) will be analyzed in the hospital biochemistry laboratory using routine methods at the beginning of the study from blood samples taken by a nurse after at least 12 hours of fasting and without consuming alcohol for 24 hours before.
Biochemical Measurements - CRP | at the beginning the study 1 times
  Participants' c-reactive protein tests (CRP) (mg/L) will be analyzed in the hospital biochemistry laboratory using routine methods at the beginning of the study from blood samples taken by a nurse after at least 12 hours of fasting and without consuming alcohol for 24 hours before.
Anthropometric Measurements - Body weight (kg) | at the beginning the study 1 times
  At the beginning and end of the study, body weights (kg) will be measured using a bioelectrical impedance (BIA) device with a sensitivity of 50 grams in accordance with the measurement standards.
Anthropometric Measurements - Height | at the beginning the study 1 times
  Height (cm) will be measured with a stadiometer in the Frankfort plane, standing and with the head upright.
Body Mass Index | at the beginning the study 1 times
  The body mass index (BMI) of the participants will calculated according to the body weight (kg) / height (m)2 formula.
Body Mass Index Classification | at the beginning the study 1 times
  The body mass index (BMI) of the participants is classified according to the World Health Organization (WHO) criteria. BMI ≤ 18.5 kg/m2 is underweight, between 18.5-24.99 kg/m2 is normal, ≥ 25 kg/m2 is overweight, and ≥ 30 kg/m2 is obese.
Anthropometric Measurements - Fat Mass | at the beginning the study 1 times
  At the beginning and end of the study, body fat mass (kg) analysis will be performed using a bioelectrical impedance (BIA) device, paying attention to measurement standards.
Anthropometric Measurements - Fat ratio calculation | at the beginning the study 1 times
  At the beginning and end of the study, body composition analyses will be performed using a bioelectrical impedance (BIA) device with measurement standards. According to the BIA analysis, fat percentage (%) will be calculated as the ratio of total body fat weight to total body weight.
Anthropometric Measurements - Fat-free mass | at the beginning the study 1 times
  At the beginning and end of the study, fat-free mass (kg) will be analyzed using a bioelectrical impedance (BIA) device, paying attention to measurement standards.
Anthropometric Measurements - Muscle mass | at the beginning the study 1 times
  At the beginning and end of the study, lean muscle mass (kg) will be analyzed using a bioelectrical impedance (BIA) device, paying attention to measurement standards.
Anthropometric Measurements - Total body water | at the beginning the study 1 times
  At the beginning and end of the study, total body water (kg) will be analyzed using a bioelectrical impedance (BIA) device, paying attention to measurement standards.
Biochemical Measurements - HbA1c | at the beginning the study 1 times
  HbA1C will be analyzed in the hospital biochemistry laboratory using routine methods from blood samples taken by a nurse at the beginning of the study.
Biochemical Measurements - Fasting Insulin | at the beginning of the study
  Fasting insulin levels (IU) will be analyzed in the hospital biochemistry laboratory using routine methods from blood samples taken by a nurse at the beginning of the study.
Biochemical Measurements - Urea | at the beginning of the study 1 times
  The blood urea (mg/dL) will be analyzed in the hospital biochemistry laboratory using routine methods from blood samples taken by a nurse at the beginning of the study.
Biochemical Measurements - Serum Albumine | at the beginning of the study 1 times
  Serum Albumine (mg/dL) will be analyzed in the hospital biochemistry laboratory using routine methods from blood samples taken by a nurse at the beginning of the study.
Biochemical Measurements - TSH | at the beginning of the study 1 times
  TSH (mUI/mL) will be analyzed in the hospital biochemistry laboratory using routine methods from blood samples taken by a nurse at the beginning of the study.
Biochemical Measurements - Free T4 | at the beginning of the study 1 times
  Free T4 (ng/dl) will be analyzed in the hospital biochemistry laboratory using routine methods from blood samples taken by a nurse at the beginning of the study.
Biochemical Measurements - Serum Electrolyte Level | at the beginning of the study 1 times
  Serum sodium, potassium and calcium (mg/dL) will be analyzed in the hospital biochemistry laboratory using routine methods from blood samples taken by a nurse at the beginning of the study.
Biochemical Measurements - Creatinine | at the beginning of the study 1 times
  Creatinine levels (mg/dL) will be analyzed in the hospital biochemistry laboratory using routine methods from blood samples taken by a nurse at the beginning of the study.
Biochemical Measurements - White blood cell (WBC) | at the beginning of the study
  The white blood cell levels (mcL) will be analyzed in the hospital biochemistry laboratory using routine methods from blood samples taken by a nurse at the beginning of the study.
Biochemical Measurements - Neutrophil count (NEU) | at the beginning of the study
  Neutrophil count (NEU) (mcL) will be analyzed in the hospital biochemistry laboratory using routine methods from blood samples taken by a nurse at the beginning of the study.
Biochemical Measurements - Platelet (PLT) | at the beginning of the study
  Neutrophil count (NEU) (mL) will be analyzed in the hospital biochemistry laboratory using routine methods from blood samples taken by a nurse at the beginning of the study.
Biochemical Measurements - Lymphocyte count (LYM) | at the beginning of the study 1 times
  Lymphocyte count (LYM) (mcL) will be analyzed in the hospital biochemistry laboratory using routine methods from blood samples taken by a nurse at the beginning of the study.
Biochemical Measurements - Systemic Immune Inflammation Index (SII) | at the beginning of the study
  Systemic Immune Inflammation Index (SII) will calculates Platelet count X Neutrophil count/Lymphocyte count.
Prognostic Inflammatory Index (PNI) | at the beginning of the study
  Prognostic Inflammatory Index (PNI) will calculated formula "10 × Serum Albumin (g/dL) + (0.005 × Total Lymphocyte Count (/mm³))".
The dietary inflammatory index | 3 days
  The dietary inflammatory index will be calculated from individuals' 24-hour food consumption averages. The dietary inflammatory index will be calculated as a total of 1,000 calories, taking into account the dietary inflammatory load of the foods consumed. In this study, the dietary inflammatory index will be calculated for a total of 27 food items.

SECONDARY OUTCOMES:
Food Consumption Record | 3 days
  The food consumption record will be taken to evaluate the nutritional status of the participants. Food consumption records will be evaluated in the BeBIS (Nutrition Information System) program and the daily energy (kcal) intake will be calculated.
Food Consumption Record | 3 days
  The food consumption record will be taken to evaluate the nutritional status of the participants. Food consumption records will be evaluated in the BeBIS (Nutrition Information System) program and the daily carbohydrate (g), protein (g), fat (g), saturated fat (g), monounsaturated fatty acid (g), polyunsaturated fatty acid (g), omega-3 fatty acids (g), omega-6 fatty acids (g), and fiber (g) intake will be calculated.
Food Consumption Record | 3 days
  The food consumption record will be taken to evaluate the nutritional status of the participants. Food consumption records will be evaluated in the BeBIS (Nutrition Information System) program and the daily vitamin E (mg), thiamine (mg), riboflavine (mg), niacin (mg), vitamine B5 (mg), vitamin B6 (mg), vitamin C, sodium (mg), potassium (mg), calcium (mg), magnesium (mg), phosphor (mg), iron (mg), zinc (mg), copper (mg), cholesterol (mg) intake will be calculated.
Bristol Stool Form Scale | at the beginning of the study
  The Bristol Stool Form Scale, developed by Lewis and Heaton in Bristol, England, is a subjective scale used to assess an individual's stool consistency and bowel habits. This scale assesses defecation status in seven groups: Type 1 and Type 2 constipation; Type 3, Type 4, and Type 5 normal defecation; and Type 6 and Type 7 diarrhea. The form will be asked to participants.
Gastrointestinal Symptom Assessment Scale | at the beginning of the study
  Developed by Revicki and colleagues and validated for Turkish by Turan et al., the GSRS is used to assess common symptoms of gastrointestinal disorders. The GSRS asks how an individual has felt about gastrointestinal issues over the past week. The scale consists of 15 questions, divided into five subscales: diarrhea (3 questions), dyspepsia (4 questions), constipation (3 questions), abdominal pain (3 questions), and reflux (2 questions). The higher the score, the more severe the gastrointestinal symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Hande Seven Avuk, Ph.D., Principal Investigator — Istanbul Bilgi University; Gökben Anıl, Principal Investigator — Haliç University
Locations (1):
- Istanbul Bilgi University, Istanbul, Uskudar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No